CLINICAL TRIAL: NCT01143571
Title: Evaluation of Skin, Colonic and Oral Microbiota and Effect of Time and Antibiotic Treatment on Organism Diversity at Each Site
Brief Title: Evaluation of Skin, Colonic, and Oral Microbiome and Effect of Time and Antibiotic Treatment on Organism Diversity at Each Site
Status: Completed | Type: Observational
Sponsor: National Cancer Institute (NCI) (NIH)
Responsible Party: Sponsor
Organization: National Institutes of Health Clinical Center (CC) (NIH)
Other Study IDs: 999910018; 10-C-N018
Record Dates: First submitted 2010-06-11; First posted 2010-06-14 (Estimated); Last update posted 2020-06-11 (Actual); Status verified 2019-06-18

CONDITIONS: BMI; General Demographics Characteristics
Keywords: Microbiome; Samples

STUDY DESIGN:
Observational Model: Ecologic or Community | Time Perspective: Prospective

SUMMARY:
Background:

* Most studies of infectious agents have focused on specific microbes, such as human papillomaviruses and cervical cancer, and the hepatitis B and C virus and liver cancer. The skin and many internal areas (including the mouth and the gastrointestinal tract) also contain large numbers of naturally occurring microbes, but these areas have not received as much study.
* Some of the infectious agents that naturally reside in the body may have an effect on health. The study of naturally occurring microbes in the human body is a new area of research, and much remains to be learned regarding the extent and pattern of their appearance and appropriate techniques for testing them.
* Researchers are interested in collecting human samples from areas known to contain naturally occurring microbes. These samples will provide baseline information for further studies.

Objectives:

- To collect a set of study samples from individuals who have applied to participate in a study assessing the relationship among the bacteria H. pylori, peptic ulcer disease, and gastric cancer.

Eligibility:

- Individuals between the ages of 21 and 65 who are participating in the clinical trial entitled A Phase III Randomized Trial of Three Antibiotic Regimens to Eradicate Helicobacter Pylori.

Design:

* Researchers will collect oral (saliva), colonic, and skin swab samples from study participants who tested positive for the presence of the H. pylori bacteria. These samples will be collected at the three study visits (enrollment, 6 weeks, and 1 year).
* Researchers will also collect samples from people who applied for the clinical trial but did not test positive for H. pylori. These samples will be collected at the enrollment visit and 1 year later.
* Blood samples will be collected at each study visit.

DETAILED DESCRIPTION:
The study of infectious agents and their role in disease is not new. Most efforts in this area have focused on specific agents, such as human papillomaviruses and cervical cancer, Helicobacter pylori (HP) and gastric diseases and carcinoma, hepatitis B and C virus and liver cancer, to name a few. The body s skin and mucosal surface s play host to microbial communities (the microbiome) whose membership outnumbers our own somatic and germ cells by an order of magnitude or more. The skin, oral, and gastrointestinal (GI) tract are all densely colonized surfaces . Recent technological advances, however, have made exploration of the microbiome, an understudied area, feasible. It is reasonable to hypothesize that some of the infectious agents that naturally reside in the body may impact health, or that perhaps the balance between the various micro-organisms has an effect on health. This new field of study has much promise that could lead to important new discoveries of how infectious agents are associated with disease and how environmental (e.g., diet) and host responses (e.g., immune response and genetics) to these agents determine chronic patterns of colonization and subsequent disease risk.

However, because the study of the human microbiome is a new area of research, much remains to be learned regarding: a) the extent and pattern of the microbiome at various sites, b) determinants of these patterns (e.g., consistency over time), and c) optimal assay techniques.

Prior to launching large-scale epidemiological studies to evaluate the association between microbiome and disease (including cancer), it is crucial to conduct well-designed, systematic, methodological studies to address some of the issues listed above. These methodological studies will begin to provide the baseline information that could be used to plan for, and conduct disease association studies.

We propose to initiate a study to collect oral, skin, vaginal (only women), penile (men only) and colonic samples at enrollment and again 6 months later on up to 150 individuals. Our objectives are:

1. To evaluate the microbiome heterogeneity between individuals across specimen types - colonic/oral/skin/vaginal/penile.
2. To evaluate the microbiome heterogeneity within individuals (over time and across specimen types - colonic/oral/skin/vaginal/penile).
3. To evaluate the effect of self-reported antibiotic treatment on the oral, colonic, skin, penile and vaginal microbiomes diversity and richness.
4. To evaluate the associations between colonic microbiome and gastrointestinal symptom disorders (assessed by the Rome III questionnaire - a detailed diagnostic questionnaire for adult functional gastrointestinal disorder), inflammatory markers (initially using measures of C-reactive protein (CRP)), and demographic factors.
5. To evaluate the reproducibility of assays used to measure the microbiota and compare the diversity and abundance determined by the different assays.

ELIGIBILITY:
* ELIGIBILITY CRITERIA:

Individuals who meet the age criteria of 18 years and older and are interested in the study will be asked to provide written informed consent. Participants must be willing to reside in the study area for the study duration (6 months). Those individuals with any known medical conditions that may limit life expectancy in the short term (including but not limited to: congestive heart failure, renal failure, prior malignancy, or any other chronic disease that limits functional status to the extent that the individual cannot perform light work or the usual activities of daily self care) are ineligible for inclusion in the study. Female participants must not be pregnant.

Individuals who report recent antibiotic use will be deferred and enrolled after they have been at least 6 weeks without antibiotic use.

In Hojancha, region of Guanacaste, Costa Rica, where our study will be conducted, a population based census was completed in March 2009 and will serve as the basis for enrollment, allowing for recruitment of a representative sample of the population. The same census was used to identify participants for another study in the same area. Therefore, because we will use the same census, we will exclude participants that were enrolled in the other study. Eligible participants must be willing to return for one follow-up visit: 6 months after the initial enrollment visit and willing to allow submission of blood for assays of serum immune markers, host genetic susceptibility and environmental factors, and to provide consent for use of the specimens.

Ages: 18 Years to 100 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: In Hojancha, region of Guanacaste, Costa Rica, where our study will be conducted, a population based census was completed in March 2009 and will serve as the basis for enrollment, allowing for recruitment of a representative sample of the population. Eligible participants must be willing to return for one follow- up visit: 6 months after the initial enrollment visit and willing to allow submission of blood for assays of serum immune markers, host genetic susceptibility and environmental factors, and to provide consent for use of the specimens. Those individuals with any known medical conditions that may limit life expectancy in the short term (including but not @@@limited to: congestive heart failure, renal failure, prior malignancy, or any other chronic disease that limits functional status to the extent that the individual cannot perform light work or the usual activities of daily self care) are ineligible for inclusion in the study. Female participants must not be pregnant.@@@
Sampling Method: Probability Sample
Enrollment: 150 (Actual)
Dates: Start 2009-11-20

PRIMARY OUTCOMES:
microbiome heterogeneity | 6 months
  To evaluate the microbiome heterogeneity between and within individuals across specimen types

CONTACTS AND LOCATIONS:
Overall Officials: Emily J Vogtmann, Ph.D., Principal Investigator — National Cancer Institute (NCI)
Locations (1):
- Proyecto Epidemiologico in Hohancha, Hojancha, Costa Rica

REFERENCES:
- [Background] Kelley JR, Duggan JM. Gastric cancer epidemiology and risk factors. J Clin Epidemiol. 2003 Jan;56(1):1-9. doi: 10.1016/s0895-4356(02)00534-6. PMID 12589864
- [Background] Parkin DM. The global health burden of infection-associated cancers in the year 2002. Int J Cancer. 2006 Jun 15;118(12):3030-44. doi: 10.1002/ijc.21731. PMID 16404738
- [Background] Peek RM Jr, Blaser MJ. Helicobacter pylori and gastrointestinal tract adenocarcinomas. Nat Rev Cancer. 2002 Jan;2(1):28-37. doi: 10.1038/nrc703. PMID 11902583